CLINICAL TRIAL: NCT00136149
Title: An Open, Prospective, Controlled Study on Immediate Placement to Evaluate Clinical Outcome of Astra Tech Implants, Fixture Microthread Osseospeed in an Immediate Loading Protocol in Extraction Sockets and Healed Ridges
Brief Title: Study on Immediate Placement to Evaluate Astra Tech Osseospeed Implants in an Immediate Loading Protocol in Extraction Sockets and Healed Ridges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/439
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immediate implants (Experimental)
  Interventions: Procedure: Immediate implants

INTERVENTIONS:
Procedure: Immediate implants — Immediate implants are used.

SUMMARY:
This is a study to evaluate immediate implants.

DETAILED DESCRIPTION:
Solitary replacement of teeth by implants in upper maxilla - immediate implants

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* Smoking
* Medical risk patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Implant survival after 1 week, 3 weeks, 8 weeks, 10 weeks, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years | after 1 week, 3 weeks, 8 weeks, 10 weeks, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be